CLINICAL TRIAL: NCT01962311
Title: Evaluation of Metabolomic Analysis in Early Diagnosis of ALS
Acronym: METABALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRN11-CA-METABALS; 2012-A00145-38 (Other: AFSSAPS)
Record Dates: First submitted 2013-01-15; First posted 2013-10-14 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: ALS
Keywords: ALS; Spinal Cerebrospinal Fluid; Urine; SERUM; Diagnosis
MeSH Terms: conditions — Disease | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): lumbar puncture
  Interventions: Procedure: lumbar puncture

INTERVENTIONS:
Procedure: lumbar puncture — lumbar puncture at enrollment in study

SUMMARY:
This project is expected to answer the question of interest assays of metabolites in the CSF as a tool for early diagnosis and should show whether it is possible or not to use such markers in the blood or urine. These studies should also help shed light on the pathophysiological original early clinical disease. While ALS appears to be more a clinical syndrome that pathophysiological entity unique metabolic abnormalities identified could help identify mechanisms disrupted in which therapeutic interventions will be possible.

DETAILED DESCRIPTION:
A blood test that would allow the diagnosis

1. to reduce the time between the first signs and diagnosis in ALS patients for therapeutic treatment earlier and
2. to exclude rapidly non ALS in their avoiding unnecessary investigations and anxiety of being infected with a terrible prognosis disease. It is currently accepted that neurodegenerative diseases such as ALS begin before the first clinical signs and the patient could benefit from a more efficient care if it was early.

Conduct a prospective study with 400 patients.

The secondary objectives are:

1. attempt to improve the predictive power of markers assays by adding new parameters
2. to check whether the assayed molecules in other environments more accessible (blood, urine) would provide equivalent diagnostic power of those assayed in the CSF
3. identify metabolic pathways disrupted early that could be related to the pathogenesis of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

* age 30-80
* Consent signed
* affiliation to a social security organism

Exclusion Criteria:

* Patients treated with RILUZOLE
* Enrollment in an other study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-02; Primary Completion 2017-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic markers studied are metabolites of cerebrospinal fluid, blood and urine measured by three complementary analytical methods | 2 years
  diagnostic criteria Diagnostic markers studied are metabolites of cerebrospinal fluid, blood and urine measured by three complementary analytical methods: GC / MS, LC / MSMS and proton NMR spectroscopy. These metabolites, the number of one hundred, can be grouped into four main groups: molecules of metabolism of carbohydrates, lipids, proteins, steroids

CONTACTS AND LOCATIONS:
Overall Officials: Christian ANDRES, MD-PHD, Study Director — University Hospital TOURS and INSERM U930
Locations (6):
- France (6):
  - Pôle Neurosciences et Spécialités ,Service de Neurologie,CHU d'Angers, Angers
  - Service de Neurologie et Pathologie du Mouvement Clinique de Neurologie, Pôle des Neurosciences et de l'Appareil Locomoteur INSERM U 837, Lille
  - Centre de Recherche de l'Institut du Cerveau et de la moëlle UPMC Paris 6,Département des Maladies du Système Nerveux, Paris
  - Service de neurologie, CHU La Milétrie, POITIERS, Faculté de Médecine, Poitiers
  - University Hospital, Strasbourg
  - CHRU -TOURS-Service de Neurologie, Tours

IPD SHARING:
Plan to Share IPD: No